CLINICAL TRIAL: NCT05877755
Title: Validation of Multi-contrast, High-resolution Cardiac Magnetic Resonance Imaging (CARDIO IRM)
Brief Title: Validation of Multi-contrast, High-resolution Cardiac Magnetic Resonance Imaging
Acronym: CARDIO-IRM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Grant Agreement ERC SMHEART (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUBX 2023/13
Record Dates: First submitted 2023-04-05; First posted 2023-05-26 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Cardiac Disease
Keywords: Cardiac MRI; Sequences; High-resolution; Multi-contrast; Imaging
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cardiac MRI acquisition (Other): 200 patients with a clinical indication for cardiac magnetic resonance imaging
  Interventions: Device: Cardiac MRI acquisition

INTERVENTIONS:
Device: Cardiac MRI acquisition — All patients will have additional images collected during the magnetic resonance imaging (MRI) examination. These are high-resolution multi-contrast cardiac MRI sequences in gradient echo or in balanced steady state free precession with synchronization on the electrocardiogram. The acquisitions last between 1 minute and 10 minutes. This duration depends on the patient's heart rate and breathing rate. The imaging protocol will last approximately 50 minutes. MRI examinations will be performed on a 1.5 Tesla clinical system with specific cardiac imaging coils.

SUMMARY:
Cardiovascular disease (CVD) causes at least 1.8 million European deaths annually, exceeding fatalities from cancer, chronic respiratory disease, and diabetes. Consequently, the fight against CVD has become the main priority of the World Health Organization. In the pursuit of understanding and treating CVD, cardiac magnetic resonance imaging (CMR) has remained the only modality capable of providing a comprehensive assessment of the heart's function and structure without harmful radiation. Unfortunately, current CMR systems remain too slow, too complex, require highly trained specialists and, as such, have presented a barrier to a wider adoption of CMR. The aim of CARDIO-IRM is to unleash the full potential of CMR to transform patient trajectories by introducing a fast, one-click, fully automated, and comprehensive imaging pipeline applicable to diagnosis, prognosis, and therapy selection in cardiology.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) causes at least 1.8 million European deaths annually, exceeding fatalities from cancer, chronic respiratory disease, and diabetes. Consequently, the fight against CVD has become the main priority of the World Health Organization. In the pursuit of understanding and treating CVD, cardiac magnetic resonance imaging (CMR) has remained the only modality capable of providing a comprehensive assessment of the heart's function and structure without harmful radiation. Unfortunately, current CMR systems remain too slow, too complex, require highly trained specialists and, as such, have presented a barrier to a wider adoption of CMR. The aim of this project is to unleash the full potential of CMR to transform patient trajectories by introducing a fast, one-click, fully automated, and comprehensive imaging pipeline applicable to diagnosis, prognosis, and therapy selection in cardiology.

This aim will be achieved by (i) creating a novel imaging technology that collects CMR data in a single continuous free-breathing scan, taking into account post-processing requirements at the very origin of CMR sequence design; (ii) exploiting the unique contrasts generated by this technology to automatically extract quantitative markers on cardiac anatomy, function, and tissue characteristics; and (iii) translating this transformative technology to a clinical setting.

This will be the first-ever integrated cardiac imaging pipeline in which CMR images are acquired in a single click, jointly represented in a single volume, and automatically analysed. This will unlock obstacles for broader acceptance of CMR and unleash the full potential of CMR to maximize its impact on patient trajectories. The results of this project will pave the way towards robust image-based strategies for personalized patient care (diagnosis, risk stratification, therapy selection, monitoring, and image-guided interventions).

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (over 18 years of age) requiring an MRI scan as part of their care.
* Male or female.
* Affiliated or beneficiary of a social security scheme
* Having given his/her oral no objection after having read the information note

Exclusion Criteria:

* Patient unable to give oral consent (guardianship, non-French speaker, etc.)
* Patient deprived of liberty
* Patient who does not meet the specific eligibility criteria for an MRI examination: pregnant women, known pathology that may interfere with acquisition (e.g. Parkinson's disease), absolute or relative contraindication to an MRI examination
* Patient participating in a therapeutic interventional trial or in a period of relative exclusion in relation to another protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2030-03-31 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
Imaging integration success | 60 months
  Measure of image quality according to signal-to-noise ratio

SECONDARY OUTCOMES:
Integration of the collected images in an internal database to develop new reconstruction and image processing algorithms specific to this application (e.g. using artificial intelligence) | 60 months
  Measure of training time and training loss function
Cardiac MRI feature: location and size of myocardial scars/fibrosis | 60 months
  Measured in mL on late gadolinium enhancement images
Cardiac MRI feature native parameter values (T1, T2, T1-rho, T2*) | 60 months
  Measured in milliseconds
CMR feature extracellular volume fraction (ECV) | 60 months
  Measured in mL/m2
CMR feature ejection fraction | 60 months
  Measured in percentage

CONTACTS AND LOCATIONS:
Overall Officials: BUSTIN Aurelien, PHD, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- Chu de Bordeaux, Pessac, France

REFERENCES:
- [Background] Bustin A, Stuber M, Sermesant M, Cochet H. Smart cardiac magnetic resonance delivering one-click and comprehensive assessment of cardiovascular disease. Eur Heart J. 2023 Feb 21;44(8):636-637. doi: 10.1093/eurheartj/ehac814. No abstract available. PMID 36638777